CLINICAL TRIAL: NCT06558357
Title: Evaluation of the Diagnostic Performance of 18-FDG PET-CT Scores for the Diagnosis of Polymyalgia Rheumatica and Comparison With Others Inflammatory Rheumatic Diseases.
Brief Title: Diagnostic Performance of 18-FDG PET-CT Scores for the Diagnosis of Polymyalgia Rheumatica
Acronym: RHUMATEP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0172 - RHUMATEP
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-06

CONDITIONS: Inflammatory Rheumatism; 18-FDG; Positron-emission Tomography
Keywords: Polymyalgia rheumatica; FDG; PET; Diagnostic performance; score
MeSH Terms: conditions — Rheumatic Fever; Polymyalgia Rheumatica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study of the diagnostic performance of 18-FDG PET scores in Polymyalgia rheumatica and comparaison with others inflammatories diseases.

DETAILED DESCRIPTION:
Polymyalgia Rheumatica is difficult to diagnostic because symptoms are non specific and many diseases can be differential diagnosis (cancer, infections, others rheumatisms...).

PET-CT is more often used to help for diagnostic of inflammatory disease, and particularly inflammatory rheumatism.

Some scores have been described to harmonize the diagnosis of Polymyalgia rheumatica.

The aim of this study is to evaluate the diagnostic performance of 18-FDG PET scores in Polymyalgia rheumatica and compared with others inflammatories diseases such as ankylosing spondylarthritis.

This is a multicentric retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* Having 18-FDG PET-CT between 2012 and 2024
* Diagnosis of inflammatory rheumatism by specialist doctor
* Adult without opposition to use there data for research
* Affiliate to social security system

Exclusion Criteria:

* Refusal participation
* Patient under juridic protection

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult with inflammatory rheumatism confirmed by specialist, with or without treatment and having a 18-FDG-PET CT.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of 18-FDG PET scores for diagnostic of Polymyalgia rheumatica. | up to 9 months
  Evaluation of the metabolism of mains joints compared to liver. Calculation of different scores described in literature.

SECONDARY OUTCOMES:
Analysis of SUV and visual fixation of mains joints. | up to 9 months
  Measure of SUV of mains joints and evaluation of the fixation compared to liver.
Diagnostic performance of 18-FDG PET scores for diagnostic of others inflammatory rheumatism. | up to 9 months
  Evaluation of the precedent scores for diagnosis of others rheumatisms. Creation of others scores if some joints seem to be interesting.
Comparaison of scores with clinical, biological and radiological data. | up to 9 months
  Search for correlation between scores and symptoms, blood test or CT/MRI exams.

CONTACTS AND LOCATIONS:
Overall Officials: Solène QUERELLOU, Study Director — CHU Brest
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement